CLINICAL TRIAL: NCT04971681
Title: Frontal-Striatal Reward Circuit Neuromodulation and Alcohol Self-Administration
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment paused when our alcohol supplier recalled and suspended manufacture of the product. When production resumed, there was not enough time remaining to successfully resume recruitment. We will examine the outcomes with the existing sample.
Sponsor: Indiana University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Susan K. Conroy, Assistant Professor of Psychiatry, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11511; P60AA007611 (NIH)
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Low frequency repetitive transcranial magnetic stimulation (rTMS) (Experimental): Low frequency repetitive transcranial magnetic stimulation (rTMS)
  Interventions: Device: Low frequency repetitive transcranial magnetic stimulation (rTMS); Device: Sham
- Sham rTMS Stimulation (Sham Comparator): Sham rTMS Stimulation
  Interventions: Device: Low frequency repetitive transcranial magnetic stimulation (rTMS); Device: Sham

INTERVENTIONS:
Device: Low frequency repetitive transcranial magnetic stimulation (rTMS) — Subjects will receive one session of low frequency repetitive transcranial magnetic stimulation (rTMS) targeting the medial prefrontal cortex (mPFC), within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 110% of motor threshold (MT), for a total of 1200 pulses
Device: Sham — The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.

SUMMARY:
This will be a single site randomized, 2-session, within-subject cross-over design pilot study. 20 enrolled (of 30 consented) subjects reporting varying levels of binge and high intensity drinking, defined as at least 2 episodes of drinking 4 (for women) or 5 (for men) drinks on an occasion over the last 5 weeks, (unless determined by PI that drinking history meets study objectives), will be enrolled. Subjects will be randomized to undergo one session of repetitive transcranial magnetic stimulation (rTMS) or sham immediately followed by the investigators rate control intravenous (IV) alcohol self-administration (ASA) paradigm. Subjects will then return 7-14 days later and undergo the same sequence of events with the opposite intervention (i.e. rTMS or sham) from session 1.

DETAILED DESCRIPTION:
This pilot study intends to address the critical unmet need to develop novel treatments for alcohol use disorder (AUD), such as repetitive transcranial magnetic stimulation (rTMS), that directly impact drinking behavior. Binge drinking and high intensity drinking, or consumption meeting at least binge criteria, is a high-risk alcohol self-administration (ASA) pattern associated with the binge-intoxication stage of AUD and the rewarding effects of alcohol. The investigators propose to quantify the impact of medial prefrontal cortex (mPFC) rTMS on ASA using the investigators novel "rate-control" paradigm. The rate control paradigm allows subjects to determine how quickly their breath alcohol concentration (BrAC) will change (increase, decrease, or stay the same) over the next 3-5 minute epoch, at the end of which brief computer-assisted assay of craving for alcohol and subjective response attributed to alcohol's effect on stimulation, sedation, liking and well-being in a manner comparable to the Brief Biphasic Alcohol Effects Scale (BAES). Each assay requires less than 20 seconds to complete and will be administered during the last ~0.5 minutes of alcohol delivery but before selection of the next rate of exposure. The ensemble provides detailed self-administered time course of alcohol exposure and corresponding time-stamped series of quantified perceptions for analysis. This approach has demonstrated sensitivity in associating self-reported high intensity drinking and the time until a binge alcohol exposure of 80 milligrams per decilitre (mg/dL).

The investigators premise is that clinically impactful neuromodulation should change ASA. Coupling rTMS to a laboratory-assessed ASA paradigm could document causal changes in drinking behavior attributable to modulation of specific neural circuits. The goal of this project is to generate preliminary data supporting the investigators central hypothesis - rTMS targeting to the mPFC, a primary cortical input to the frontal-striatal reward (FSR) circuit, will decrease the rate of alcohol self-administration.

ELIGIBILITY:
Inclusion Criteria:

1. Overtly healthy men and women aged 21 - 35
2. Able to give informed consent
3. Able to understand/complete questionnaires and procedures in English
4. Willing and able to adhere to the study schedule
5. At least 2 binge drinking events (at least 4 or 5 drinks on a drinking day for women and men respectively over the last 5 weeks, unless determined by study physicians that drinking history meets study objectives
6. Have venous access sufficient to allow blood sampling

Exclusion Criteria:

1. Pregnant or breast-feeding
2. Desire to be treated for any substance use disorder or court ordered to not drink alcohol
3. Medical disorders or other conditions, such as lifetime history of a seizure, including history of Electroconvulsive therapy (ECT) but excluding febrile seizures and those induced by substance withdrawal, that may influence study outcome or subject safety
4. First degree relative with idiopathic epilepsy or other seizure disorder
5. Diagnostic and Statistical Manual (DSM) 5 Disorders (non-AUD) or current/history of neurological disease of cerebral origin, or head injury with > 20 min loss of consciousness, if determined by the study physicians to affect subject safety or data integrity
6. Positive urine drug screen for amphetamines/ methamphetamines, barbiturates, benzodiazepines, cocaine, opiates, or phencyclidine if determined by the study physicians to adversely affect subject safety or data integrity
7. Medications (past 30 days) that could influence subject data/subject safety (e.g. antidepressants, antipsychotics, benzodiazepines, etc.) as determined by study physicians
8. Positive BrAC reading at beginning of any study session
9. Actively suicidal (for example, any suicide attempts within the past 3 months or any current suicidal intent, including a plan) or are at serious suicidal risk, by clinical judgment of the study physicians
10. Any condition for which the study physicians determine it is unsafe or not prudent to enroll a subject

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Conroy, MD, Principal Investigator — Indiana University
Locations (1):
- Neural Systems Lab, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy men and women were recruited from past participants consented to be contacted for future studies, through flyers placed on public bulletin boards, and through ads placed in a local emailed jobs list. Minimum criteria included age 21-35 and consumption of at least 4 drinks/day on at least 2 days in a recent 35 day period
Groups:
- Active rTMS Condition First, Then Sham rTMS: Subjects will undergo 2 sessions, one active rTMS, one sham, one week apart.
  Active session: subjects will receive low frequency repetitive transcranial magnetic stimulation (rTMS) targeting the medial prefrontal cortex (mPFC). The stimulus will consist of a continuous 20-minute train of 1 Hz rTMS, at 110% of motor threshold (MT), for a total of 1200 pulses.
- Sham rTMS Stimulation, Then Active rTMS: Subjects will undergo 2 sessions, one active rTMS, one sham, one week apart.
  Sham session: All procedures identical except that rTMS will not be delivered. The sham treatment mimics cutaneous stimulation, facilitating double-blinding.
Period: First Intervention
Arm/Group | Active rTMS Condition First, Then Sham rTMS | Sham rTMS Stimulation, Then Active rTMS
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0
Period: Washout (7-14 Days)
Arm/Group | Active rTMS Condition First, Then Sham rTMS | Sham rTMS Stimulation, Then Active rTMS
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Active rTMS Condition First, Then Sham rTMS | Sham rTMS Stimulation, Then Active rTMS
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0
Period: Followup
Arm/Group | Active rTMS Condition First, Then Sham rTMS | Sham rTMS Stimulation, Then Active rTMS
Started | 4 | 5
Completed | 3 | 5
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Within-subjects design, all subjects participated in both arms of the study
Groups:
- Active rTMS First: Subjects counterbalanced to session order Active rTMS-Sham rTMS
- Sham rTMS First: Subjects counterbalanced to order Sham rTMS-Active rTMS
- Total: Total of all reporting groups
Arm/Group | Active rTMS First | Sham rTMS First | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Customized [Count of Participants; unit: Participants] — Limited to 21-35 years old
  Participants
    Age 21-35 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 4 | 2 | 6
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: T80
Description: The amount of time subjects take to self-administer enough alcohol to raise their breath alcohol concentration (BrAC) to 80 mg/dL
Time Frame: 90 min
Measure: Mean (Standard Error); unit: Minutes
Groups:
- Low Frequency Repetitive Transcranial Magnetic Stimulation (rTMS): Subjects will receive one session of low frequency repetitive transcranial magnetic stimulation (rTMS) targeting the medial prefrontal cortex (mPFC), within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 110% of motor threshold (MT), for a total of 1200 pulses. Session order is counterbalanced.
- Sham rTMS Stimulation: Subjects will receive one session of sham stimulation. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding. Session order is counterbalanced.
Arm/Group | Low Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) | Sham rTMS Stimulation
Number analyzed (Participants) | 9 | 9
Minutes | 61.5 (9.4) | 71.6 (8.0)
Statistical Analysis 1: Comparison: Low Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) vs Sham rTMS Stimulation; Test type: Superiority; p < 0.27, t-test, 2 sided

2. Secondary Outcome: Alcohol Consumption (Drinks/Week)
Description: Alcohol consumption as measured by Time Line Follow Back (TLFB) comparing drinking baseline (5 weeks prior to study) with post-treatment during the 5-week follow-up period. The Timeline Follow-back (TLFB) is uses a calendar to assess a subject's retrospective estimates of their daily drinking.
Time Frame: 5 weeks
Measure: Mean (Standard Error); unit: Drinks/week
Arm/Group | Low Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) | Sham rTMS Stimulation
Number analyzed (Participants) | 8 | 8
Drinks/week | 14.8 (4.9) | 7.8 (3.5)
Statistical Analysis 1: Comparison: Low Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) vs Sham rTMS Stimulation; Test type: Superiority; p < 0.10, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 7 - 14 days (interval from start of Session 1 day to end of Session 2 day)
Arm/Group | Low Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) | Sham rTMS Stimulation
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT04971681/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT04971681/ICF_000.pdf